CLINICAL TRIAL: NCT05306483
Title: Transcatheter Versus Surgical Closure of Ventricular Septal Defect: A Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MS97/2021
Record Dates: First submitted 2022-03-10; First posted 2022-04-01 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2020-06

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital

STUDY DESIGN:
Intervention Model Description: The population of our intervention study is divided into two groups of participants receive different interventions.
  group (A) Patients undergoing surgical VSD closure (control group) group (B) Patients undergoing transcatheter VSD closure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventricular septal defect closure surgery (Active Comparator): Surgical closure would be done under general anesthesia, hypothermic cardiopulmonary bypass and cardioplegic arrest. Chest would be opened through standard median sternotomy Surgical techniques would be determined according to the nature of every defect and includes direct closure, patch closure which involves the use of autologous pericardium; however, polyethylene terephthalate (Dacron; C.R Bard, Haverhill, MA) and expanded polytetrafluoroethylene (Gore-Tex; W.L. Gore & Associates, Inc.,AZ) may be occasionally used. These patches are held with continuous or interrupted sutures. Direct closure (without a patch may be done for the very small defects.Most VSDs would be repaired through right atriotomy to avoid the the undesirable effects of the trans ventricular approach.
  Interventions: Procedure: Ventricular septal defect closure surgery
- catheter closure of ventricular septal defect (Active Comparator): Under general anesthesia, patients will be fully heparinized (100IU/Kg) with follow up by activated clotting time. IntraoperativeTEE will be done for more detailed assessment of the defect size, relation to the surrounding structures especially the distance from the tricuspid and the aortic valve to guide the procedure and for proper assessment after device positioning yet before its release.
  Left ventricular angiogram will be done in LAO 60, cranial 30 projection to define location and size of the defect. Accordingly, proper selection of the device siz.
  Interventions: Procedure: Ventricular septal defect closure catheter

INTERVENTIONS:
Procedure: Ventricular septal defect closure surgery — Ventricular septal defect closure surgery
  Other Names: patients undergoing surgical VSD closure
  Arms: Ventricular septal defect closure surgery
Procedure: Ventricular septal defect closure catheter — Catheter closure of VSD
  Other Names: Patients undergoing VSD trans catheter
  Arms: catheter closure of ventricular septal defect

SUMMARY:
The aim of this study is to compare Safety, efiicacy and clinical effects of surgical versus transcatheter closure of ventricular septal defect (VSD ).

The outcome of interest is success rate, residual shunts, effect on tricuspid and aortic valves, need for blood transfusion, length of hospital and intensive care unit ( ICU ) stay, complications especially complete heart block, affection of kidney functions due to the procedure length caused by Cardiopulmonary bypass in case of surgical group or by the dye used in the group of transcatheter closure.

DETAILED DESCRIPTION:
Both of transcatheter and surgical closure of VSD is a well-established procedure. Despite the wide using of both procedures, there is a defect in the evidence comparing the short-term outcome and the value of both techniques. Our multicenter study aims to compare the immediate outcome of both procedures in Egypt.

1. INTRODUCTION/ REVIEW with variable degrees of successes. Perimembranous VSDs have more intensiveLock et al in 1988 . Ventricular septal defects are the most common congenital heart diseases in children and are the second most common congenital abnormality in adults(1). nearly accounting for one-third of all cases. The extent of the opening may vary from the pin size to complete absence of the ventricular septum. There are 4 main types of VSD, the most common one of them is membranous type which accounts for almost 80% of all VSDs (2). Most isolated muscular and perimembranous VSDs (pm VSDs) are small and close spontaneously. Large eccentric pmVSDs were recommended to be closed for fear of infective endocarditis, aortic regurgitation, and pulmonary hypertension(3). Surgical closure is still considered the gold standard management since being first reported in 1955(4). However, transcatheter closure of some types of VSDs has been introduced into the clinical practice as an alternative to the surgical repair. Transcatheter closure of VSDs were initially made with the occluders of atrial septal defect (ASD) & patent ductus arteriosus (PDA) as reported by Lock in 1988 (5) with variable degrees of successes. Perimembranous VSD have more intensive demands on device design due to their nearness to the aortic valve. Hijazi et al. were first to report a successful closure of perimembranous defects with the occluder in six patients.(6) AMPLATZER muscular VSD occluder still the most common used device for transcatheter closure of muscular VSDs with generally accepted results.(7) However, The high cost of catheter closure, as well as device-related complications such as complete heart block (CHB), device embolization, aortic and tricuspid valves regurgitation, had limited its use (8) . nonetheless, the outcomes of using the transcatheter procedure to treat Perimembranous ( pm) VSD have been improved significantly in recent years because of improvement in device design and operator skills (9).

   Superiority of one procedure over the other is still an issue of debate. Consecutively, it is now possible to compare the outcome of both techniques as the data comparing the outcome of them are so limited.
2. METHODOLOGY:

   Patients and Methods/ Subjects and Methods/ Material and Methods. Type of Study: Prospective purposed comparative study.
3. Study setting:

   The study will be conducted at both of Academic institute of cardiac surgery and National Heart Institute.

   Study Period: One year. Start point: Once the protocol approved from the ethical committee.

   Study Population:

   The population of study is divided into two groups, Patients undergoing surgical VSD closure group(control group) & Patients undergoing catheter VSD closure group.
4. Patient evaluation & selection:

   All patients will be evaluated by independent cardiologist.
5. Sampling Method Patients who are suitable for transcatheter closure according to the Indian guidelines 2019 will be offered transcatheter closure firstly, other eligible cases for the study but not suitable for transcatheter closure or patients who have any troubles with transcatheter closure, will be treated surgically.

Sample Size:

72 patients divided into 36 patients in each group using pass 2 program for sample size calculation according to previous literature(12). setting power at 80%, α error at 0.05.

6. Ethical Considerations:

All the following will be applied:

* Informed consent will be taken.
* Patient information sheet will be given to the patients. - Confidentiality & Privacy.
* Privileged communication.
* Respect and responsibility.

  7. Study Procedures: An informed consent would be taken from the parents of the patients. All procedures would be performed under general anesthesia.

Note: my role is only to observe and assist only.Each patient in both groups would be subjected to:

* Full history taking.
* General examination.
* Cardiac examination.
* Routine investigations which include 12 lead ECG, Laboratory investigations (CBC, PT, PTT, ESR, CRP, Urea, Creatinine, liver enzymes, bilirubin), Chest X-ray P/A view.
* Complete diagnostic transthoracic examination by 2D ECHO, doppler and color flow mapping with probe frequencies appropriate for each patient size to assess:

I. Interatrial septum. II. Interventricular septal defects (number, size and site). III. Left Ventricle dimensions, volume and systolic function. IV. All cardiac valves morphology and flow. V. Right ventricle size &systolic function by TAPSE. VI. Estimated Right ventricular systolic pressure (RVSP ) using tricuspid regurgitation (TR) jet and/or estimated mean pulmonary artery pressure (PAP) using PR regurgitation jet.

▪ Surgical closure of VSD: Surgical closure would be done under general anesthesia, hypothermic cardiopulmonary bypass and cardioplegic arrest. Chest would be opened through standard median sternotomy (13). Surgical techniques would be determined according to the nature of every defect and includes direct closure, patch closure which involves. All patients will be transferred to the ICU for further follow up and management.

▪ Transcatheter closure of VSD: done for more detailed assessment of the defect size, to guide the procedure and for proper assessment after device positioning yet before its release. the use of autologous pericardium; however, polyethylene terephthalate (Dacron; C.R Bard, Haverhill, MA) and expanded polytetrafluoroethylene (Gore-Tex; W.L. Gore & Associates, Inc., AZ) may be occasionally used. These patches are held with continuous or interrupted sutures. Direct closure (without a patch may be done for the very small defects14. Most VSDs would be repaired through right atriotomy to avoid the undesirable effects of ventriculostomies(14). Under general anesthesia, patients will be fully heparinized (100 IU/Kg) with follow up by activated clotting time. Intraoperative TEE will be relation to the surrounding structures especially the distance from the tricuspid and the aortic valves

Left ventricular angiogram will be done in left anterior oblique (LAO ) 60 degree , cranial 30 degree projection to define location and size of the defect. Accordingly, proper selection of the device size(15) . Only FDA approved devices would be used, after release of the device left ventricular angiography will assure proper device positioning, and transoesophageal (TEE ) or trans thoracic echocardiograph(TTE) will be used to assess nearby structures and nearby valvular flow.

All the patients will recover from the general anesthesia, then transmitted to the ICU for follow up.

The patients of each group will have all the routine labs repeated, 12 leads electrocardiogram (ECG), complete TTE and chest x-ray, all these data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Ventricular septal defect: All patients who have congenital VSD which require intervention and accepting the selected measure of intervention. Surgery closure for Perimembranous VSD which is not suitable for catheter closure, muscular VSD. Catheter closure for Perimembranous VSD with at least 4 mm distal from aortic valve, mid muscular, anterior muscular.
* Age: Pediatric age group with minimum age of 10 months to 18 years old.
* Gender: both males and females.
* Intervention classification: Elective.
* NYHA classification: I - III
* weight more than 8 Kg.
* left to right shunt with Qp/Qs more than 1.5.

Exclusion Criteria:

* Non-congenital VSD.
* severe pulmonary hypertension with right to left shunt.
* ischemic stroke
* hemorrhage stroke
* systemic thromboembolism
* heart failure
* rheumatic heart disease
* cardiac valvular abnormalities
* infective endocarditis
* high degree atrioventricular block
* atrial fibrillation, atrial flutter
* paroxysmal supraventricular tachycardia
* endocardial cushing syndome,
* Ebstein's anomaly
* hemodynamically significant atrial septal defect
* transposition of great vessels
* tetralogy of Fallot.

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 72 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Rate of Transthoracic Echocardiography residual ventricular septal defect shunts | One year
  two-dimensional Transthoracic Echocardiography for Detection of persistent residual Ventricular septal defect shunt flow - physiological parameter

SECONDARY OUTCOMES:
Incidence of Transthoracic Echocardiography tricuspid and aortic valves regurgitation detect | One year
  Transthoracic Echocardiography detection of change or damage in tricuspid or aortic valve - physiological parameter
% of patients with need for blood transfusion | One week postoperative
  Bleeding
length of hospital or ICU stay | One month
  Postoperative complaints need more hospital or ICU stay
Rate of Electrocardiogram complete heart block | One month
  Electrocardiogram ECG to detect type of heart block and degree of the damage to conducting pathways - physiological parameter

CONTACTS AND LOCATIONS:
Locations (1):
- Hamdy Singab, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be shared. Results will be published by the investigators in academic journals

REFERENCES:
- [Result] Hoffman JI, Kaplan S. The incidence of congenital heart disease. J Am Coll Cardiol. 2002 Jun 19;39(12):1890-900. doi: 10.1016/s0735-1097(02)01886-7. PMID 12084585
- [Result] Alahmadi MH, Oliver TI. Ventricular Septal Defect. 2024 Oct 16. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK470330/ PMID 29261884
- [Result] Mongeon FP, Burkhart HM, Ammash NM, Dearani JA, Li Z, Warnes CA, Connolly HM. Indications and outcomes of surgical closure of ventricular septal defect in adults. JACC Cardiovasc Interv. 2010 Mar;3(3):290-7. doi: 10.1016/j.jcin.2009.12.007. PMID 20298987
- [Result] LILLEHEI CW, COHEN M, WARDEN HE, VARCO RL. The direct-vision intracardiac correction of congenital anomalies by controlled cross circulation; results in thirty-two patients with ventricular septal defects, tetralogy of Fallot, and atrioventricularis communis defects. Surgery. 1955 Jul;38(1):11-29. No abstract available. PMID 14396676
- [Result] Lock JE, Block PC, McKay RG, Baim DS, Keane JF. Transcatheter closure of ventricular septal defects. Circulation. 1988 Aug;78(2):361-8. doi: 10.1161/01.cir.78.2.361. PMID 3396173
- [Result] Hijazi ZM, Hakim F, Haweleh AA, Madani A, Tarawna W, Hiari A, Cao QL. Catheter closure of perimembranous ventricular septal defects using the new Amplatzer membranous VSD occluder: initial clinical experience. Catheter Cardiovasc Interv. 2002 Aug;56(4):508-15. doi: 10.1002/ccd.10292. PMID 12124963
- [Result] Holzer R, Balzer D, Cao QL, Lock K, Hijazi ZM; Amplatzer Muscular Ventricular Septal Defect Investigators. Device closure of muscular ventricular septal defects using the Amplatzer muscular ventricular septal defect occluder: immediate and mid-term results of a U.S. registry. J Am Coll Cardiol. 2004 Apr 7;43(7):1257-63. doi: 10.1016/j.jacc.2003.10.047. PMID 15063439
- [Result] Sullivan ID. Transcatheter closure of perimembranous ventricular septal defect: is the risk of heart block too high a price? Heart. 2007 Mar;93(3):284-6. doi: 10.1136/hrt.2006.103671. Epub 2006 Oct 11. PMID 17035508
- [Result] Masura J, Gao W, Gavora P, Sun K, Zhou AQ, Jiang S, Ting-Liang L, Wang Y. Percutaneous closure of perimembranous ventricular septal defects with the eccentric Amplatzer device: multicenter follow-up study. Pediatr Cardiol. 2005 May-Jun;26(3):216-9. doi: 10.1007/s00246-005-1003-7. PMID 16082578
- [Result] Saxena A, Relan J, Agarwal R, Awasthy N, Azad S, Chakrabarty M, Dagar KS, Devagourou V, Dharan BS, Gupta SK, Iyer KS, Jayranganath M, Joshi R, Kannan B, Katewa A, Kohli V, Kothari SS, Krishnamoorthy KM, Kulkarni S, Kumar RM, Kumar RK, Maheshwari S, Manohar K, Marwah A, Mishra S, Mohanty SR, Murthy KS, Rao KN, Suresh PV, Radhakrishnan S, Rajashekar P, Ramakrishnan S, Rao N, Rao SG, Chinnaswamy Reddy HM, Sharma R, Shivaprakash K, Subramanyan R, Kumar RS, Talwar S, Tomar M, Verma S, Vijaykumar R. Indian guidelines for indications and timing of intervention for common congenital heart diseases: Revised and updated consensus statement of the Working group on management of congenital heart diseases. Ann Pediatr Cardiol. 2019 Sep-Dec;12(3):254-286. doi: 10.4103/apc.APC_32_19. PMID 31516283
- [Result] Kouchoukos NT, Blackstone EH, Kirklin JW. Surgical implications of pulmonary hypertension in congenital heart disease. Adv Cardiol. 1978;(22):225-31. doi: 10.1159/000401033. PMID 619518
- [Result] JULIAN OC, LOPEZ-BELIO M, DYE WS, JAVID H, GROVE WJ. The median sternal incision in intracardiac surgery with extracorporeal circulation; a general evaluation of its use in heart surgery. Surgery. 1957 Oct;42(4):753-61. No abstract available. PMID 13467646
- [Result] Merrick AF, Lal M, Anderson RH, Shore DF. Management of ventricular septal defect: a survey of practice in the United Kingdom. Ann Thorac Surg. 1999 Sep;68(3):983-8. doi: 10.1016/s0003-4975(99)00689-x. PMID 10509995
- [Result] Odemis E, Saygi M, Guzeltas A, Tanidir IC, Ergul Y, Ozyilmaz I, Bakir I. Transcatheter closure of perimembranous ventricular septal defects using Nit-Occlud((R)) Le VSD coil: early and mid-term results. Pediatr Cardiol. 2014 Jun;35(5):817-23. doi: 10.1007/s00246-013-0860-8. Epub 2014 Jan 12. PMID 24413836
- See also: Faculty of medicine, Ain shams university,cairo, Egypt — http://med.asu.edu.eg